CLINICAL TRIAL: NCT06112665
Title: ToFAcitinib in Early Active Axial SpondyloarThritis: a Prospective, Randomized, Double-BLind, PlAcebo-CoNtrolled MulticEntre Study
Brief Title: ToFAcitinib in Early Active Axial SpondyloarThritis:
Acronym: FASTLANE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Denis Poddubnyy, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FASTLANE1
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: This is a phase IV, multicentre, randomized, double-blind, placebo-controlled study designed to compare the efficacy and safety of tofacitinib versus placebo (on a background of an NSAID) over 16 weeks of treatment and 4 weeks of safety follow-up in subjects with early active axSpA and inadequate response to at least one NSAID, with objective signs of inflammation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: multicentre, randomized, double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofactinib (Experimental): Patients receive Tofacitinib and Naproxene
  Interventions: Drug: Tofacitinib 5 MG
- Placebo Arm (Active Comparator): Patients receive placebo pills and Naproxene
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — Patients receive Tofacitinib and Naproxene

SUMMARY:
This is a phase IV, multicentre, randomized, double-blind, placebo-controlled study designed to compare the efficacy and safety of tofacitinib versus placebo (on a background of an NSAID) over 16 weeks of treatment and 4 weeks of safety follow-up in subjects with early active axSpA and inadequate response to at least one NSAID, with objective signs of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of axSpA and fulfilment of the ASAS classification criteria
* Symptom (back pain) duration for ≤ 2 years, according to the definition of early axial SpA by ASAS.
* Active disease activity as defined by: BASDAI ≥4 and back pain score (BASDAI question 2) of ≥4 AND objective signs of inflammation evident by osteitis in MRI of SIJ AND/OR elevated serum CRP levels.

Exclusion criteria:

* active current infection, severe infections in the last 3 months
* history of recurrent Herpes zoster or disseminated Herpes simplex
* immunodeficiency
* chronic Hepatitis B, C or HIV infection
* women: pregnant or lactating (have to practice reliable method of contraception)
* other severe diseases conflicting with a clinical study, contraindications for MRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Main trial endpoint | 16 weeks
  Proportion of subjects achieving disease remission defined as Ankylosing Spondylitis Disease Activity Score (ASDAS)CRP<1.3 at week 16 from baseline

SECONDARY OUTCOMES:
Change from baseline in the MRI SIJ SPARCC osteitis score at week 16 | 16 weeks
  Change from baseline in the MRI SIJ SPARCC osteitis score at week 16

CONTACTS AND LOCATIONS:
Overall Officials: Denis Poddubbnyy, Prof. Dr. med., Principal Investigator — Charité Rheumatology
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after study enrollment end
Access Criteria: not known yet

REFERENCES:
- [Derived] Rios Rodriguez V, Sanchez-Riera L, Haibel H, Hoppner C, Torgutalp M, Proft F, Rademacher J, Binder E, Diehl A, Vranic I, Zhao Y, Mundayat R, Yndestad A, Poddubnyy D. Tofacitinib in early active axial spondyloarthritis: protocol of a randomized double-blind, placebo-controlled, multicenter phase IV study, FASTLANE. Ther Adv Musculoskelet Dis. 2025 Mar 12;17:1759720X251324429. doi: 10.1177/1759720X251324429. eCollection 2025. PMID 40078463